CLINICAL TRIAL: NCT02891226
Title: A Phase 2, Multicenter, Randomized, Parallel-Arm, Placebo-Controlled Study of LY3074828 in Subjects With Active Crohn's Disease (SERENITY)
Brief Title: A Study of Mirikizumab (LY3074828) in Participants With Active Crohn's Disease
Acronym: SERENITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16492; I6T-MC-AMAG (Other: Eli Lilly and Company); 2016-002204-84 (EudraCT Number)
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Results first posted 2022-02-28 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Crohn's Disease
Keywords: inflammatory bowel disease; IL-23; biologic
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — mirikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirikizumab (Experimental): Period 1 (Weeks 0 -12): 200 Milligram (mg), 600 mg, and 1000 mg mirikizumab administered intravenously (IV) every 4 Weeks (Q4W).
  Period 2 (Weeks 12 - 52): 200 mg, 600 mg, and 1000 mg mirikizumab administered IV Q4W; 300 mg mirikizumab administered subcutaneously (SC) Q4W; 1000 mg mirikizumab administered IV Q4W for non-improvers in period 1; and 1000 mg mirikizumab administered IV Q4W for participants on placebo during period 1.
  Period 3 (Weeks 52 - 208): 300 mg mirikizumab administered SC Q4W.
  Interventions: Drug: Mirikizumab
- Placebo (Placebo Comparator): Period 1 (Weeks 0 -12): Participants received placebo administered intravenously (IV) Q4W.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirikizumab
  Other Names: LY3074828
  Arms: Mirikizumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the study drug Mirikizumab in participants with active Crohn's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Active Crohn's Disease (CD) as determined by the SES-CD, and participant reported stool frequency and abdominal pain.
* Inadequate response or failure to tolerate at least one of the following: aminosalicylates; budesonide; systemic corticosteroids; immunosuppressants (eg, azathioprine, 6-mercaptopurine, or methotrexate); or prior exposure to biologics for the treatment of CD.

Exclusion Criteria:

* Have complications of CD such as strictures, stenoses, or any other manifestation for which surgery might be indicated, or that could confound the evaluation of efficacy.
* Diagnosis of conditions affecting the digestive tract, such as ulcerative colitis, indeterminate colitis, fistulizing disease, abdominal or perianal abscess, adenomatous colonic polyps not excised, colonic mucosal dysplasia, and short bowel syndrome.
* Have had any kind of bowel resection, diversion, or placement of a stoma within 6 months or any other intra-abdominal surgery within 3 months prior to screening.
* Are unsuitable for inclusion in the study in the opinion of the investigator or sponsor for any reason that may compromise the subject's safety or confound data interpretation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2016-12-14 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2021-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (108):
- United States (44):
  - Longwood Research, Huntsville, Alabama
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Valley View Internal Medicine, Garden Grove, California
  - Ventura Clinical Trials, Ventura, California
  - Delta Waves Sleep Disorders and Research Center, Colorado Springs, Colorado
  - Medical Research Center of Connecticut, Hamden, Connecticut
  - Clinical Research of West Florida, Clearwater, Florida
  - Wellness Clinical Research, Hialeah Gardens, Florida
  - University of Miami, Miami, Florida
  - Vista Health Research, Miami, Florida
  - Clinical Neuroscience Solutions Inc, Orlando, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - Robley Rex VAMC, Louisville, Kentucky
  - Health Quest Medical Care, Owensboro, Kentucky
  - Delta Research Partners LLC, Monroe, Louisiana
  - Louisiana Research Center, Shreveport, Louisiana
  - MedStar Health Research Institute, Rosedale, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - Huron Gastroenterology Associates, Ypsilanti, Michigan
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - Las Vegas Medical Research, Las Vegas, Nevada
  - Holy Name Medical Center, Teaneck, New Jersey
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Consultants For Clinical Research, Cincinnati, Ohio
  - University Hospitals Health Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Healthcare Research Consultant, Tulsa, Oklahoma
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Gastro One, Germantown, Tennessee
  - Advanced Gastroenterology, Union City, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Hermann Drive Surgical Hospital, Houston, Texas
  - Digestive Health Associates of Texas, Richardson, Texas
  - San Antonio Gastroenterology, San Antonio, Texas
  - Care Access Research - Salt Lake City, Salt Lake City, Utah
  - Virginia Mason Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
- Australia (4):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Ballarat Health Services - Base Hospital, Ballarat, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
- Belgium (2):
  - Hospital Universitaire Erasme Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Sudbury Endoscopy Centre, Greater Sudbury, Ontario, Canada
- Czechia (6):
  - Krajska zdravotni a.s. - Masarykova nemocnice v Usti nad Labem, o.z., Ústí nad Labem, Czech Republic
  - Hepato-gastroenterologie HK, s.r.o., Hradec Králové
  - Gregar s.r.o., Olomouc
  - Fakultni Nemocnice v Motole, Prague
  - Thomayerova Nemocnice, Praha 4 - Krc
  - Krajska nemocnice T. Bati a.s., Zlín
- Hungary (2):
  - Obudai Egeszsegugyi Centrum Kft, Budapest
  - Javorszky Odon Hospital, Vác
- Japan (13):
  - Toho University School of Medicine, Sakura Hospital, Sakura-shi, Chiba
  - Kitakyushu Municipal Medical Center, Kitakyusyu-shi, Fukoka
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Hokkaido P.W.F.A.C. Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Sameshima Hospital, Kagoshima, Kagoshima-ken
  - Gokeikai Ofuna Chuo Hospital, Kamakura-shi, Kanagawa
  - Takagi Clinic, Sendai, Miyagi
  - Kinshukai Infusion Clinic, Osaka, Osaka
  - Tokyo Medical And Dental University Hospital, Bunkyo-ku, Tokyo
  - Kyorin University Hospital, Mitaka, Tokyo
  - JHCO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo
  - Toyama Prefectural Central Hospital, Toyama, Toyama
  - Fukuoka University Hospital, Fukuoka
- Netherlands (4):
  - St Elisabeth Ziekenhuis, Tilburg, North Brabant
  - Academisch Medisch Centrum, Amsterdam
  - Radboud Universitair Medisch Centrum Nijmegen, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (7):
  - Szpital Uniwersytecki nr 2 im. dr J. Biziela, Bydgoszcz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - SOLUMED Centrum Medyczne, Poznan
  - Korczowski Bartosz, Gabinet Lekarski, Rzeszów
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia Matki, Dziecka i Mlodziezy, Warsaw
  - Melita Medical Sp. Z O. O., Wroclaw
- Romania (3):
  - SC Pelican SRL, Oradea, Bihor County
  - SC Med Life SA, Bucharest
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Russia (11):
  - Novosibirsk State Medical University, Novosibirsk
  - FSBI Scientific Research Inst. of Physyology and Basic Medic, Novosibirsk
  - Ultramed, Omsk
  - City Clinical Hospital # 2 n.a. Fedor Khristoforovich Gral, Perm
  - Private Medical Institution Evromedservis, Pushkin
  - Baltic Medicine, Saint Petersburg
  - City Hospital of Saint Martyr Elizabeth, Saint Petersburg
  - LLC Scientific Research Centre EKO-Bezopasnost, Saint Petersburg
  - Medical Institute REAVIZ, Samara
  - NonState Healthcare Institution Central Clinical Hospital, Samara
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
- Universitätsspital Zürich, Zurich, Switzerland
- Ukraine (9):
  - Kyiv Municipal Clinical Hospital #1, Kyiv
  - Communal institution of the Kyiv Regional Council "Kyiv Regional Clinical Oncology Dispensary", Kyiv
  - Lviv Regional Central Hospital, Lviv
  - Odesa Regional Clinical Hospital, Odesa
  - A. Novak Transcarpathian Regional Clinical Hospital, Uzhhorod
  - Vinnitsa City Clinical Hospital #1, Vinnytsia
  - SRI of Invalid Rehabil.,Educ.Scient.Med.Complex, Vinnytsia
  - City Clinical Hospital #6, Zaporizhzhia
  - CI City Hospital #1, Zaporizhzhia
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Magro F, Protic M, De Hertogh G, Chan LS, Pollack P, Jairath V, Carlier H, Hon E, Feagan BG, Harpaz N, Pai R, Reinisch W. Effects of Mirikizumab on Histologic Resolution of Crohn's Disease in a Randomized Controlled Phase 2 Trial. Clin Gastroenterol Hepatol. 2024 Sep;22(9):1878-1888.e10. doi: 10.1016/j.cgh.2023.11.010. Epub 2023 Nov 20. PMID 37993033
- [Derived] Sands BE, Peyrin-Biroulet L, Kierkus J, Higgins PDR, Fischer M, Jairath V, Hirai F, D'Haens G, Belin RM, Miller D, Gomez-Valderas E, Naegeli AN, Tuttle JL, Pollack PF, Sandborn WJ. Efficacy and Safety of Mirikizumab in a Randomized Phase 2 Study of Patients With Crohn's Disease. Gastroenterology. 2022 Feb;162(2):495-508. doi: 10.1053/j.gastro.2021.10.050. Epub 2021 Nov 5. PMID 34748774
- See also: A Study of Mirikizumab (LY3074828) in Participants With Active Crohn's Disease (SERENITY) — https://trials.lillytrialguide.com/en-US/trial/5IDfzP6WruCqkOq0OokSSe

RESULTS

PARTICIPANT FLOW:
Groups:
- Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W): Participants received placebo administered intravenously (IV) Q4W.
- Period 1: 200 Milligram (mg) Mirikizumab IV Q4W: Participants received 200 mg mirikizumab administered IV Q4W.
- Period 1: 600 mg Mirikizumab IV Q4W: Participants received 600 mg mirikizumab administered IV Q4W.
- Period 1: 1000 mg Mirikizumab IV Q4W: Participants received 1000 mg mirikizumab administered IV Q4W.
- Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers): Participants received 200 mg mirikizumab administered IV Q4W. Participants improved on the same mirikizumab dose in Period 1.
- Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers): Participants received 600 mg mirikizumab administered IV Q4W. Participants improved on the same mirikizumab dose in Period 1.
- Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers): Participants received 1000 mg mirikizumab administered IV Q4W. Participants improved on the same mirikizumab dose in Period 1.
- Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers): Participants received 300 mg mirikizumab administered SC Q4W. Participants improved on any mirikizumab dose in Period 1.
- Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers): Participants who did not improve in Period 1 on mirikizumab (any dose) received 1000 mg mirikizumab administered IV Q4W.
- Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo): Participants who received placebo in period 1 received 1000 mg mirikizumab administered IV Q4W.
- Period 3: 300 mg Mirikizumab SC Q4W: Participants received 300 mg mirikizumab administered SC Q4W.
- Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2: Participants did not receive drug during the follow-up period. Group includes participants who received 200 mg mirikizumab IV Q4W during period 2.
- Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers): Participants did not receive drug during the follow-up period. Group includes participants who received 1000 mg mirikizumab IV Q4W during period 2 after improving on the same dose in Period 1.
- Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers): Participants did not receive drug during the follow-up period. Group includes participants who did not improve in period 1, and received 1000 mg mirikizumab IV Q4W during period 2.
- Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1): Participants did not receive drug during the follow-up period. Group includes participants who received placebo in period 1 and 1000 mg mirikizumab administered IV Q4W.
- Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3: Participants did not receive drug during the follow-up period. Group includes participants who received 300 mg mirikizumab administered SC Q4W during period 3.
Period: Period 1 (Weeks 0 to 12)
Arm/Group | Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W) | Period 1: 200 Milligram (mg) Mirikizumab IV Q4W | Period 1: 600 mg Mirikizumab IV Q4W | Period 1: 1000 mg Mirikizumab IV Q4W | Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers) | Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo) | Period 3: 300 mg Mirikizumab SC Q4W | Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2 | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers) | Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1) | Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3
Started | 64 | 31 | 32 | 64 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least 1 Dose of Study Drug | 64 | 31 | 32 | 64 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 59 | 29 | 28 | 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 2 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Enrollment Failure | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Weeks 12 to 52)
Arm/Group | Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W) | Period 1: 200 Milligram (mg) Mirikizumab IV Q4W | Period 1: 600 mg Mirikizumab IV Q4W | Period 1: 1000 mg Mirikizumab IV Q4W | Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers) | Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo) | Period 3: 300 mg Mirikizumab SC Q4W | Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2 | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers) | Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1) | Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3
Started | 0 (Participants were assigned to this arm during period 1.) | 0 (Participants were assigned to this arm during period 1.) | 0 (Participants were assigned to this arm during period 1.) | 0 (Participants were assigned to this arm during period 1.) | 9 (Participants were assigned to this arm during period 2.) | 9 (Participants were assigned to this arm during period 2.) | 23 (Participants were assigned to this arm during period 2.) | 46 (Participants were assigned to this arm during period 2.) | 30 (Participants were assigned to this arm during period 2.) | 59 (Participants were assigned to this arm during period 2.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 8 | 8 | 20 | 41 | 24 | 42 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 5 | 6 | 17 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PI decision due to Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PI and Sponsor Decision due to Subject Safety | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PI Decision due to Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Endoscopic Procedure was not Evaluated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy and Withdrew from Study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3 (Weeks 52 to 208)
Arm/Group | Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W) | Period 1: 200 Milligram (mg) Mirikizumab IV Q4W | Period 1: 600 mg Mirikizumab IV Q4W | Period 1: 1000 mg Mirikizumab IV Q4W | Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers) | Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo) | Period 3: 300 mg Mirikizumab SC Q4W | Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2 | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers) | Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1) | Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3
Started | 0 | 0 | 0 | 0 | 0 (Participants were assigned to this arm during period 2.) | 0 (Participants were assigned to this arm during period 2.) | 0 (Participants were assigned to this arm during period 2.) | 0 (Participants were assigned to this arm during period 2.) | 0 (Participants were assigned to this arm during period 2.) | 0 (Participants were assigned to this arm during period 2.) | 137 (Participants were assigned to this arm during period 3.) | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 137 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 0 | 0 | 0 | 0 | 0
Not completed — Roll over to AMAX | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 108 | 0 | 0 | 0 | 0 | 0
Not completed — Decided to not Participate in Extension Period (Week 104-208) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — PI Decision as Subject Not Responding to Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance With Study Visit Schedule | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W) | Period 1: 200 Milligram (mg) Mirikizumab IV Q4W | Period 1: 600 mg Mirikizumab IV Q4W | Period 1: 1000 mg Mirikizumab IV Q4W | Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers) | Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo) | Period 3: 300 mg Mirikizumab SC Q4W | Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2 | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers) | Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1) | Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 (Participants were assigned to this arm during follow-up period.) | 2 (Participants were assigned to this arm during follow-up period.) | 1 (Participants were assigned to this arm during follow-up period.) | 1 (Participants were assigned to this arm during follow-up period.) | 3 (Participants were assigned to this arm during follow-up period.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Placebo IV Q4W: Participants received placebo administered IV Q4W.
- 200 mg Mirikizumab IV Q4W: Participants received 200 mg mirikizumab administered IV Q4W.
- 600 mg Mirikizumab IV Q4W: Participants received 600 mg mirikizumab administered IV Q4W.
- 1000 mg Mirikizumab IV Q4W: Participants received 1000 mg mirikizumab administered IV Q4W.
- Total: Total of all reporting groups
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W | Total
Number analyzed (Participants) | 64 | 31 | 32 | 64 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.00 (13.04) | 38.10 (11.80) | 40.40 (13.33) | 37.70 (13.11) | 38.70 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 14 | 18 | 30 | 98
  Male | 28 | 17 | 14 | 34 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 2 | 2 | 8
  Not Hispanic or Latino | 53 | 27 | 26 | 54 | 160
  Unknown or Not Reported | 7 | 4 | 4 | 8 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 7 | 1 | 4 | 8 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 3 | 4 | 11
  White | 55 | 28 | 24 | 52 | 159
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 3 | 0 | 0 | 1 | 4
  Belgium | 0 | 1 | 1 | 4 | 6
  Czechia | 4 | 1 | 0 | 5 | 10
  Hungary | 3 | 1 | 0 | 3 | 7
  Japan | 6 | 1 | 4 | 7 | 18
  Netherlands | 2 | 3 | 0 | 2 | 7
  Poland | 6 | 6 | 3 | 9 | 24
  Romania | 0 | 0 | 1 | 4 | 5
  Russia | 6 | 3 | 2 | 3 | 14
  Ukraine | 4 | 5 | 4 | 6 | 19
  United Kingdom | 1 | 0 | 0 | 0 | 1
  United States | 29 | 10 | 17 | 20 | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Endoscopic Response at Week 12
Description: Endoscopic response defined as ≥ 50% reduction from baseline in Simple Endoscopic Score for Crohn's Disease (SES-CD) at Week 12. The SES-CD evaluates 4 endoscopic variables: presence and size of ulcers, proportion of surface covered by ulcers, proportion of surface affected by disease, and presence and severity of stenosis. The total SES-CD calculated as sum of 4 variables for 5 bowel segments: (ileum;right,transverse,and left colon;and rectum): presence and size of ulcers (none = score 0; diameter 0.1-0.5 cm = score 1; 0.5-2 cm = score 2; >2 cm = score 3); extent of ulcerated surface (none = 0; <10% = 1;10-30% = 2;>30% = 3);extent of affected surface (none = 0; <50% = 1;50-75% = 2;>75% =3); and presence and type of narrowings (none=0; single, can be passed=1; multiple,can be passed=2; cannot be passed=3). Total SES-CD scores range from 0 to 56, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: All randomized participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 64 | 31 | 32 | 64
percentage of participants | 10.9 [4.5 to 17.4] | 25.8 [12.9 to 38.7] | 37.5 [23.4 to 51.6] | 43.8 [33.6 to 53.9]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.079, Regression, Logistic; Odds Ratio (OR) = 2.75, 90% CI 2-sided [1.07 to 7.08]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.003, Regression, Logistic; Odds Ratio (OR) = 4.92, 90% CI 2-sided [2.01 to 12.07]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 6.14, 90% CI 2-sided [2.81 to 13.42]

2. Secondary Outcome: Percentage of Participants Achieving Endoscopic Remission at Week 12
Description: Endoscopic remission defined as SES-CD of <4 ileal-colonic or <2 for isolated ileal disease, and no subscore >1 at week 12. The SES-CD evaluates 4 endoscopic variables: presence and size of ulcers, proportion of surface covered by ulcers, proportion of surface affected by disease, and presence and severity of stenosis. The total SES-CD is calculated as the sum of the 4 variables for the 5 bowel segments: (ileum; right, transverse, and left colon; and rectum): presence and size of ulcers (none = score 0; diameter 0.1-0.5 cm = score 1; 0.5-2 cm = score 2; greater than (>) 2 cm = score 3); extent of ulcerated surface (none = 0; less than (<) 10% = 1; 10-30% = 2; >30% = 3); extent of affected surface (none = 0; <50% = 1; 50-75% = 2; >75% = 3); and presence and type of narrowings (none=0; single, can be passed=1; multiple, can be passed=2; cannot be passed=3). Total SES-CD scores range from 0 to 56, with higher scores indicating more severe disease.
Time Frame: Week 12
Population: All randomized participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 64 | 31 | 32 | 64
percentage of participants | 1.6 [0.0 to 4.1] | 6.5 [0.0 to 13.7] | 15.6 [5.1 to 26.2] | 20.3 [12.0 to 28.6]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.241, Regression, Logistic; Odds Ratio (OR) = 4.31, 90% CI 2-sided [0.55 to 33.58]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.032, Regression, Logistic; Odds Ratio (OR) = 11.16, 90% CI 2-sided [1.76 to 70.64]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.009, Regression, Logistic; Odds Ratio (OR) = 16.04, 90% CI 2-sided [2.82 to 91.32]

3. Secondary Outcome: Percentage of Participants Achieving Patient Reported Outcome Remission at Week 12
Description: PRO remission is defined as stool frequency (SF) ≤2.5 and abdominal pain (AP) ≤1 and no worse than baseline at week 12. SF captures the number of liquid or very soft stools. AP score is classified as 0=none, 1=mild, 2=moderate, 3=severe.
Time Frame: Week 12
Population: All randomized participants.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 64 | 31 | 32 | 64
percentage of participants | 6.3 [1.3 to 11.2] | 12.9 [3.0 to 22.8] | 28.1 [15.1 to 41.2] | 21.9 [13.4 to 30.4]
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.330, Regression, Logistic; Odds Ratio (OR) = 2.0, 90% CI 2-sided [0.62 to 6.45]
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.006, Regression, Logistic; Odds Ratio (OR) = 5.72, 90% CI 2-sided [2.02 to 16.21]
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.029, Regression, Logistic; Odds Ratio (OR) = 3.52, 90% CI 2-sided [1.37 to 9.07]

4. Secondary Outcome: Mean Change From Baseline on the Patient Global Rating - Severity (PGRS) Crohn's Disease Score at Week 12
Description: The PGRS is a 1-item patient-rated questionnaire designed to assess the participant's rating of their disease symptom severity over the past 24 hours. Responses are graded on a 6-point scale in which a score of 1 indicates the subject has no symptoms (that is, "none") and a score of 6 indicates that the participant's symptom are "very severe." Least Squares Mean (LS Mean) was calculated using Mixed Model for Repeated Measures (MMRM) model with treatment, geographic region, geographic region, prior biologic CD therapy use (prior biologic experience versus prior biologic naive), baseline score, visit, and the interaction of treatment-by-visit and baseline-by-visit as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who had a baseline and at least one post-baseline PGRS value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 58 | 26 | 29 | 56
score on a scale | -0.44 (0.132) | -1.08 (0.194) | -1.27 (0.189) | -0.98 (0.134)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.007, Mixed Models Analysis; LS Mean difference (Final Values) = -0.64, 90% CI 2-sided [-1.03 to -0.25], Standard Error of Mean 0.234
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = -0.83, 90% CI 2-sided [-1.21 to -0.45], Standard Error of Mean 0.230
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.005, Mixed Models Analysis; LS Mean difference (Final Values) = -0.53, 90% CI 2-sided [-0.84 to -0.22], Standard Error of Mean 0.188

5. Secondary Outcome: Mean of Patient Global Rating - Change (PGRC) Crohn's Disease Score at Week 12
Description: The PGRC scale is a patient-rated instrument designed to assess the participant's rating of change in their symptom(s). Responses are graded on a 7-point Likert scale in which a score of 1 indicates that the participant's symptom is "very much better," a score of 4 indicates that the participant's symptom has experienced "no change," and a score of 7 indicates that the participant's symptom is "very much worse."
Time Frame: Baseline, Week 12
Population: All randomized participants who had a baseline and at least one post-baseline PGRC value.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 56 | 29 | 27 | 57
score on a scale | 3.6 (1.11) | 2.8 (1.26) | 2.6 (0.97) | 2.5 (0.89)

6. Secondary Outcome: Mean Change From Baseline on the Inflammatory Bowel Disease Questionnaire (IBDQ) Score at Week 12
Description: The IBDQ is a 32-item self-administered questionnaire. The IBDQ has 4 dimensions: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items), and social function (5 items). Responses are graded on a 7-point Likert scale in which 7 denotes "not a problem at all" and 1 denotes "a very severe problem." Scores range from 32 to 224; a higher score indicates a better quality of life. LS Mean was calculated using Mixed Model for Repeated Measures (MMRM) model with treatment, geographic region, geographic region, prior biologic CD therapy use (prior biologic experience versus prior biologic naive), baseline score, visit, and the interaction of treatment-by-visit and baseline-by-visit as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who had a baseline and at least one post-baseline IBDQ value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 56 | 29 | 28 | 57
score on a scale | 17.11 (3.725) | 41.16 (5.311) | 46.57 (5.244) | 42.35 (3.770)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = 24.05, 90% CI 2-sided [13.53 to 34.56], Standard Error of Mean 6.358
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = 29.46, 90% CI 2-sided [18.84 to 40.08], Standard Error of Mean 6.421
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = 25.24, 90% CI 2-sided [16.67 to 33.82], Standard Error of Mean 5.185

7. Secondary Outcome: Mean Change From Baseline on the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Score at Week 12
Description: The Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Scale is a13-item, symptom-specific questionnaire that specifically assesses the participant's self-reported severity of fatigue and its impact upon daily activities and functioning. The FACIT-F uses a numeric rating scale of 0-4 associated with a range over "Not at all" to "Very much" for each item to assess fatigue and its impact in the past 7 days. Total scores range from 0 to 52, with higher scores indicating less fatigue. LS Mean was calculated using Mixed Model for Repeated Measures (MMRM) model with treatment, geographic region, geographic region, prior biologic CD therapy use (prior biologic experience versus prior biologic naive), baseline score, visit, and the interaction of treatment-by-visit and baseline-by-visit as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who had a baseline and at least one post-baseline FACIT-F value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 56 | 29 | 28 | 57
score on a scale | 2.90 (1.209) | 10.81 (1.728) | 9.09 (1.721) | 9.62 (1.223)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = 7.91, 90% CI 2-sided [4.48 to 11.34], Standard Error of Mean 2.072
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Test type: Superiority; p = 0.004, Mixed Models Analysis; LS Mean difference (Final Values) = 6.20, 90% CI 2-sided [2.72 to 9.67], Standard Error of Mean 2.102
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = 6.73, 90% CI 2-sided [3.94 to 9.51], Standard Error of Mean 1.686

8. Secondary Outcome: Mean Change From Baseline on the 36-Item Short Form Health Survey (SF-36) Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores at Week 12
Description: The SF-36 is a health-related survey that assesses participant's quality of life and consists of 36 questions covering 8 health domains:physical functioning, bodily pain, role limitations due to physical problems and emotional problems, general health, mental health, social functioning, vitality, 2 component scores (MCS and PCS). MCS consisted of social functioning, vitality, mental health, and role-emotional scales. PCS consisted of physical functioning, bodily pain, role-physical, and general health scales. Each domain is scored by summing individual items and transforming scores into a 0 to 100 scale with higher scores indicating better health status or functioning. LS Mean was calculated using Mixed Model for Repeated Measures (MMRM) model with treatment, geographic region, geographic region, prior biologic CD therapy use (prior biologic experience versus prior biologic naive), baseline score, visit, and the interaction of treatment-by-visit and baseline-by-visit as fixed factors.
Time Frame: Baseline, Week 12
Population: All randomized participants who had a baseline and at least one post-baseline PCS and MCS value.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo IV Q4W | 200 mg Mirikizumab IV Q4W | 600 mg Mirikizumab IV Q4W | 1000 mg Mirikizumab IV Q4W
Number analyzed (Participants) | 56 | 29 | 28 | 57
score on a scale
  MCS | 2.34 (1.133) | 7.47 (1.602) | 6.52 (1.592) | 6.05 (1.152)
  PCS | 3.11 (0.774) | 4.70 (1.096) | 8.01 (1.108) | 6.70 (0.787)
Statistical Analysis 1: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Mental Component Summary (MCS); Test type: Superiority; p = 0.008, Mixed Models Analysis; LS Mean difference (Final Values) = 5.14, 90% CI 2-sided [1.95 to 8.32], Standard Error of Mean 1.927
Statistical Analysis 2: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Mental Component Summary (MCS); Test type: Superiority; p = 0.033, Mixed Models Analysis; LS Mean difference (Final Values) = 4.18, 90% CI 2-sided [0.96 to 7.41], Standard Error of Mean 1.951
Statistical Analysis 3: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Mental Component Summary (MCS); Test type: Superiority; p = 0.021, Mixed Models Analysis; LS Mean difference (Final Values) = 3.71, 90% CI 2-sided [1.08 to 6.34], Standard Error of Mean 1.589
Statistical Analysis 4: Comparison: Placebo IV Q4W vs 200 mg Mirikizumab IV Q4W; Physical Component Summary (PCS); Test type: Superiority; p = 0.229, Mixed Models Analysis; LS Mean difference (Final Values) = 1.59, 90% CI 2-sided [-0.59 to 3.77], Standard Error of Mean 1.319
Statistical Analysis 5: Comparison: Placebo IV Q4W vs 600 mg Mirikizumab IV Q4W; Physical Component Summary (PCS); Test type: Superiority; p < 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = 4.91, 90% CI 2-sided [2.67 to 7.14], Standard Error of Mean 1.349
Statistical Analysis 6: Comparison: Placebo IV Q4W vs 1000 mg Mirikizumab IV Q4W; Physical Component Summary (PCS); Test type: Superiority; p = 0.001, Mixed Models Analysis; LS Mean difference (Final Values) = 3.60, 90% CI 2-sided [1.81 to 5.38], Standard Error of Mean 1.078

9. Secondary Outcome: Population Pharmacokinetics (PopPK): Mean Population Clearance of Mirikizumab
Description: Population mean (between-subject coefficient variance [CV %]) apparent clearance. Clearance is estimated based on concentration data collected in the time frame of 0-208 weeks.
Time Frame: Week 0, 4, 8: Predose, end of infusion; Week 2; 4; 6; 8, 11-12; 12-13; 16; 20; 24; 28; 36; 44; 52; 60; 68; 76; 84; 92; 104; 108; 112; 120; 128; 136; 144; 156; 164; 172; 180; 188; 196 and 208 weeks post infusion
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per Hour (L/h)
Groups:
- Mirikizumab IV Q4W: Participants received 200 mg, 600 mg, 1000 mg mirikizumab administered IV Q4W.
Arm/Group | Mirikizumab IV Q4W
Number analyzed (Participants) | 186
Liters per Hour (L/h) | 0.0225 (30)

10. Secondary Outcome: Population Pharmacokinetics (PopPK): Mean Population Volume of Distribution of Mirikizumab
Description: Population mean (between-subject coefficient variance [CV %]) apparent volume of distribution. Volume of distribution is estimated based on concentration data collected in the time frame of 0-208 weeks.
Time Frame: as for outcome 9
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters (L)
Arm/Group | Mirikizumab IV Q4W
Number analyzed (Participants) | 186
Liters (L) | 5.05 (18)

ADVERSE EVENTS:
Time Frame: Baseline Up To 208 Weeks
Description: All randomized participants who received at least 1 dose of study drug. Gender specific events occurring only in male or female participants have had the number of participants at risk adjusted accordingly.
Arm/Group | Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W) | Period 1: 200 Milligram (mg) Mirikizumab IV Q4W | Period 1: 600 mg Mirikizumab IV Q4W | Period 1: 1000 mg Mirikizumab IV Q4W | Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) | Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers) | Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo) | Period 3: 300 mg Mirikizumab SC Q4W | Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2 | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers) | Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1) | Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/31 | 0/32 | 0/64 | 0/9 | 0/9 | 0/23 | 0/46 | 0/30 | 0/59 | 0/136 | 0/1 | 0/2 | 0/1 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 7/64 | 0/31 | 3/32 | 2/64 | 0/9 | 0/9 | 0/23 | 2/46 | 3/30 | 9/59 | 15/136 | 0/1 | 0/2 | 0/1 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 24/64 | 11/31 | 12/32 | 27/64 | 7/9 | 5/9 | 14/23 | 30/46 | 16/30 | 30/59 | 89/136 | 0/1 | 1/2 | 1/1 | 0/1 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W) (N=64) | Period 1: 200 Milligram (mg) Mirikizumab IV Q4W (N=31) | Period 1: 600 mg Mirikizumab IV Q4W (N=32) | Period 1: 1000 mg Mirikizumab IV Q4W (N=64) | Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) (N=9) | Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) (N=9) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) (N=23) | Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers) (N=46) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers) (N=30) | Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo) (N=59) | Period 3: 300 mg Mirikizumab SC Q4W (N=136) | Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2 (N=1) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers) (N=2) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers) (N=1) | Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1) (N=1) | Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3 (N=3)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Maternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/36 (0) | 0/14 (0) | 0/18 (0) | 0/30 (0) | 0/4 (0) | 0/4 (0) | 0/12 (0) | 0/23 (0) | 1/13 (1) | 0/33 (0) | 0/61 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0/1 (0)
Paternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0/28 (0) | 0/17 (0) | 0/14 (0) | 0/34 (0) | 0/5 (0) | 0/5 (0) | 0/11 (0) | 0/23 (0) | 0/17 (0) | 0/26 (0) | 2/75 (2) | 0/0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/2 (0)
Blood potassium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/36 (0) | 0/14 (0) | 0/18 (0) | 0/30 (0) | 0/4 (0) | 0/4 (0) | 0/12 (0) | 0/23 (0) | 1/13 (1) | 0/33 (0) | 0/61 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0/1 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Period 1: Placebo Intravenous (IV) Every 4 Weeks (Q4W) (N=64) | Period 1: 200 Milligram (mg) Mirikizumab IV Q4W (N=31) | Period 1: 600 mg Mirikizumab IV Q4W (N=32) | Period 1: 1000 mg Mirikizumab IV Q4W (N=64) | Period 2: 200 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) (N=9) | Period 2: 600 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) (N=9) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Improvers) (N=23) | Period 2: 300mg Mirikizumab Subcutaneous (SC) Q4W (Period 1 Mirikizumab Improvers) (N=46) | Period 2: 1000 mg Mirikizumab IV Q4W (Period 1 Mirikizumab Non-improvers) (N=30) | Period 2: 1000 mg Mirkizumab IV Q4W (Period 1 Placebo) (N=59) | Period 3: 300 mg Mirikizumab SC Q4W (N=136) | Follow-up Period: 200 mg Mirikizumab IV Q4W in Period 2 (N=1) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Improvers) (N=2) | Follow-up Period: 1000 mg Mirikizumab IV Q4W in Period 2 (Period 1 Mirikizumab Non-improvers) (N=1) | Follow-up Period: 1000 mg Mirkizumab IV Q4W in Period 2 (Placebo in Period 1) (N=1) | Follow-up Period: 300 mg Mirikizumab SC Q4W in Period 3 (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 2 (2) | 5 (6) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 8 (10) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (15) | 1 (1) | 4 (64) | 1 (7) | 3 (16) | 8 (162) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 18 (114) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0/28 (0) | 0/17 (0) | 0/14 (0) | 0/34 (0) | 0/5 (0) | 0/5 (0) | 1/11 (2) | 0/23 (0) | 0/17 (0) | 0/26 (0) | 0/75 (0) | 0/0 (0) | 0 (0) | 0/0 (0) | 0/0 (0) | 0/2 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human anaplasmosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 6 (7) | 3 (3) | 4 (6) | 25 (33) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 5 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 2 (2) | 3 (3) | 14 (18) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 1/36 (1) | 0/14 (0) | 0/18 (0) | 0/30 (0) | 0/4 (0) | 1/4 (1) | 0/12 (0) | 0/23 (0) | 0/13 (0) | 2/33 (2) | 2/61 (2) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0/1 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 8 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 2 (4) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 6 (6) | 1 (1) | 3 (4) | 8 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 2 (3) | 7 (7) | 0 (0) | 0 (0) | 3 (4) | 4 (4) | 3 (4) | 4 (4) | 16 (30) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0/36 (0) | 0/14 (0) | 0/18 (0) | 0/30 (0) | 0/4 (0) | 0/4 (0) | 1/12 (1) | 0/23 (0) | 0/13 (0) | 0/33 (0) | 0/61 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0/1 (0)
Endometriosis (Reproductive system and breast disorders) | 0/36 (0) | 0/14 (0) | 0/18 (0) | 0/30 (0) | 0/4 (0) | 0/4 (0) | 1/12 (1) | 0/23 (0) | 0/13 (0) | 0/33 (0) | 0/61 (0) | 0 (0) | 0/0 (0) | 0 (0) | 0 (0) | 0/1 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 11 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 5 years from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02891226/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/26/NCT02891226/SAP_001.pdf